CLINICAL TRIAL: NCT04020445
Title: Simplification of Complex Insulin Regimens With Preserving Good Glycemic Control in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Bekes County Central Hospital (Other)
Collaborators: University of Debrecen (Other); Szeged University (Other)
Responsible Party: Principal Investigator, Zoltán Taybani, Principal investigator, Bekes County Central Hospital
Other Study IDs: BekesCCH
Record Dates: First submitted 2019-07-10; First posted 2019-07-16 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: HBA1c; Body Weight; Hypoglycemia
Keywords: iDegLira; deintensification; overtreatment; simplification; type 2 diabetes
MeSH Terms: conditions — Body Weight; Hypoglycemia; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: de-escalation of complex insulin regimens — complex insulin regimens are switched to fix ratio combinations consisting of of a basal insulin and a GLP-1 (glucagon-like peptide-1) receptor agonist

SUMMARY:
This study examines prospectively the safety and efficacy of switching from multiple daily insulin injections (MDI) to once daily IDegLira (insulin degludec and liraglutide fix ratio combination), a fixed-ratio combination of insulin degludec and liraglutide, in relatively well controlled (HbA1c<7.5%) subjects with type 2 diabetes using low total daily insulin dose (TDD).

DETAILED DESCRIPTION:
Type 2 diabetic patients suffering from severe hyperglycemia are often apply multiple daily insulin injections (MDI). If glucose toxicity resolves, the regimen may potentially be simplified, but there are no specific guidelines regarding this and a lot of patients are left on MDI.

The Investigators aimed to examine prospectively the safety and efficacy of switching from MDI to once daily IDegLira, a fixed-ratio combination of insulin degludec and liraglutide, in relatively well controlled (HbA1c<7.5%) subjects with type 2 diabetes using low total daily insulin dose (TDD).

The investigators hypothesize that in everyday clinical practice switching from low dose MDI to IDegLira in patients of different ages with well-controlled (or overcontrolled) type 2 diabetes is safe, may induce weight loss and result in similar or better glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic (T2D) patients >18 years old
* detectable random, non-fasting serum C-peptide levels
* HbA1c=< 7.5%
* treated with MDI (with stable daily doses of insulin at least for 90 days prior to baseline visit)
* using relatively low total daily insulin dose (TDD), at baseline visit low TDD is defined as TDD<70 IU/day and TDD<0.6 IU/kg/day at the same time.

Exclusion Criteria:

* Type 1 diabetes
* treatment of T2D with any medication for diabetes other than insulin or metformin during 90 days before baseline visit
* active cancer
* anaemia (haemoglobin <100g/l)
* acute or chronic kidney disease with an estimated glomerular filtration rate <30 mL/min/1.73 m2

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Well-controlled or overtreated adult type 2 diabetic patients using relatively low dose MDI.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Number of participants reaching HbA1c<7% and HbA1c<6.5% | it is checked at baseline and at 3, 6, 9 and 12 months
  HbA1c is measuerd by laboratory blood test
change in body weight from baseline to 3, 6, 9 and 12 months | it is checked at baseline and at 3, 6, 9 and 12 months
  body weight is measured at the diabetes ambulance
change in risk of hypoglycemia from baseline to 3, 6, 9 and 12 months | it is checked at baseline and at 3, 6, 9 and 12 months
  hypoglycemia risk is assessed by analysing the patients' diary

CONTACTS AND LOCATIONS:
Overall Officials: Zoltán J Taybani, MD, Principal Investigator — Bekes County Central Hospital
Locations (1):
- Zoltán Taybani, Békéscsaba, Bekes County, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Taybani Z, Botyik B, Katko M, Gyimesi A, Varkonyi T. Simplifying Complex Insulin Regimens While Preserving Good Glycemic Control in Type 2 Diabetes. Diabetes Ther. 2019 Oct;10(5):1869-1878. doi: 10.1007/s13300-019-0673-8. Epub 2019 Jul 25. PMID 31347100